CLINICAL TRIAL: NCT05846672
Title: Turkish Cultural Adaptation, Validity, and Reliability of the "Gait Outcomes Assessment List for Children With Lower-Limb Difference Parent Version/ Child Version" in Pediatric Rheumatologic Diseases
Brief Title: Turkish Cultural Adaptation, Validity and Reliability of the "Gait Outcomes Assessment List"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc. Prof., Istanbul University - Cerrahpasa
Other Study IDs: NAAAArman
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Rheumatologic Disease; Pediatric ALL; Children, Only; Lower Extremity Problem
MeSH Terms: conditions — Collagen Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ultimate goal of treating children with lower extremity differences is to improve quality of life, optimize function, and maximize participation by addressing the physical, social, and psychological effects of lower extremity differences. In the pediatric field, research has focused on the Body Functions and Structures area of the ICF framework, such as radiographic measurements of limb alignment and length, postoperative complications, and recovery time. Priority targets for children/parents are better captured in the Activity and Participation areas of the ICF framework.

Developed in Canada, the Gait Outcomes Assessment List (GOAL)was created to evaluate outcomes for gait-related interventions for children with cerebral palsy based on a wide range of children's and parents' goals. It was also developed for other childhood conditions associated with lower extremity disorders. The present study aimed to determine the Turkish cultural adaptation, validity, and reliability of the "Gait Outcomes Assessment List for Children With Lower-Limb Difference Parent Version/ Child Version" in Pediatric Rheumatologic Diseases.

DETAILED DESCRIPTION:
The International Classification of Functioning, Disability, and Health (ICF) is a useful framework for assessing and categorizing lower extremity problems. The ultimate goal of treating children with lower extremity differences is to improve quality of life, optimize function, and maximize participation by addressing the physical, social, and psychological effects of lower extremity differences. Research on this topic in the pediatric field has focused on the Body Functions and Structures area of the ICF framework, such as radiographic measurements of limb alignment and length, postoperative complications, and recovery time. While this area is an important predictor of the technical success of an intervention, it cannot be assumed that these are priority targets for children/parents. It also does not correspond to the most important factor in quality of life outcomes. Priority targets are better captured in the Activity and Participation areas of the ICF framework.

Gait Outcomes Assessment List (GOAL) is a multidimensional, self-administered child and parent report developed using the Priority Framework as its conceptual framework.

Developed in Canada, the GOAL was created to evaluate outcomes for gait-related interventions for children with cerebral palsy based on a wide range of children's and parents' goals. It was also developed for other childhood conditions associated with lower extremity disorders. Lower extremity and walking functions change due to joint swelling, effusion, tenderness, and painful restriction in joint movement, which are common, especially in load-bearing joints in pediatric rheumatological diseases. These changes affect kinematic and kinetic parameters and cause functional limitations. Evaluation of functional limitations within the framework of ICF, especially within the scope of participation, forms the basis of "treat-to-target" conception.

The present study was designed to determine the Turkish cultural adaptation, validity, and reliability of the "Gait Outcomes Assessment List for Children With Lower-Limb Difference Parent Version/ Child Version" in Pediatric Rheumatologic Diseases. To evaluate the validity, Childhood Health Assessment Questionnaire (CHAQ), Six Minute Walk Test (6MWT), and 10 Stair Climb Test (10SCT) will be applied. The Turkish form of GOAL will be applied again after 7 days to evaluate reliability. All forms will be applied by a physiotherapist.

This study plans to include 200 children with chronic rheumatological disease. Factor analysis methods will be used in the analysis of the factor structure of the scale, and correlation analyses (Pearson and Spearman coefficients) will be used in the analysis of validity and test-retest reliability. Cronbach's alpha analysis will be used in the reliability analysis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Diagnosed with chronic rheumatological disease
* 6-18 ages
* Have reading and writing skills
* Residing in Turkey
* To have the cognitive skills to understand and answer the questions in the questionnaires

Exclusion Criteria:

* Have had lower extremity surgery in the past 6 months
* Have had lower extremity surgery in the past 6 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosed with pediatric rheumatological disease aged 6-18 years, treated in the pediatric rheumatology clinic of Istanbul University Medical Faculty Hospital and who meet the inclusion criteria will be included in our study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Gait Outcomes Assessment List for Children with Lower-Limb Difference (GOAL-LD) | Change from baseline to 7 day
  It was developed by Dermott et al. The original version of the parent- and child-reported GOAL questionnaire used in this study, consists of 44 items across seven domains: (A) Walking and getting around, (B) Pain/Discomfort/Fatigue, (C) Physical Activities, Games & Recreation, (D) Gait Appearance, (E) Use of Braces & Assistive Devices, and (F) Body Image & Self-Esteem.
6 Minute Walk Test (6 MWT) | Baseline
  The 6-minute walk test is a well-tolerated, easy-to-apply and simple test that shows the submaximal level of functional capacity. This test measures the distance that participants can walk quickly on a hard and flat surface in 6 minutes. Participants rest in a chair near the starting position for at least 10 minutes before the start of the test. Before and after the test, heart rate, blood pressure, saturation are measured, and fatigue level is determined with the Modified Borg scale. Participants are told how to perform the test. At the end of the test, the distance walked by the participants in 6 minutes will be recorded in meters.
10 Stair Climb Test (10SCT) | Baseline
  10 Stair Climb Test is a measure of ability to ascend and descend a flight of stairs. We will ask the patient to go walk as quickly as patients feel safe and comfortable to the top of the 10 stairs, and than turn around, and come back down. Physiotherapist will stop the clock when the patients second foot touches the landing. Seconds will recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc. Prof., Principal Investigator — Istanbul University-Cerrahpaşa, Faculty of Health Science; Asena Yekdaneh, Pt. MSc., Study Chair — Fenerbahce University; Asya Albayrak, Pt. MSc., Study Chair — Istanbul Kent University; Nuray Aktay Ayaz, Prof. Dr., Study Chair — Istanbul University Medical Faculty; Ayşenur Namlı, Pt. MSc., Study Chair — Aydın University; Fatma Gül Demirkan, MD, Study Chair — Istanbul University Medical Faculty; Özlem Akgün, MD, Study Chair — Istanbul University Medical Faculty
Locations (1):
- Istanbul University Medical Faculty Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No